CLINICAL TRIAL: NCT06475391
Title: The Effects of L-arginine Supplementation on Anaerobic Exercise Performance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: HE2024-0063
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Skeletal Muscle; Human Performance
MeSH Terms: interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-arginine (Experimental): Participants will ingest 2 grams of L-arginine before completing three anaerobic exercise tasks (grip strength, vertical jump, and Wingate cycle ergometer test).
  Interventions: Dietary Supplement: L-arginine
- Placebo (Placebo Comparator): Participants will ingest 2 grams of placebo (dextrose) before completing three anaerobic exercise tasks (grip strength, vertical jump, and Wingate cycle ergometer test).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L-arginine — 2 grams iof L-arginine will be ingested before an acute testing bout of exercise tasks in 250 mL of cranberry juice.
  Arms: L-arginine
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate if acute ingestion of L-arginine will enhance anaerobic exercise performance in young, healthy, and recreationally active adults.

DETAILED DESCRIPTION:
After being enrolled in the study you will be measured on a number of parameters including: body circumferences, body composition via bioelectrical impedance analysis (BIA), height, weight, resting blood pressure, and resting heart rate.

All participants will be asked to complete the same protocol for this study. The study design is a randomized, double-blind, placebo controlled, cross-over type of study. What this means is that each participant in the study will complete two exercise sessions after ingesting either a placebo (dextrose - a sugar molecule) or the active ingredient [insert supplement] plus dextrose. Neither you nor the research assistant testing you on the exercise sessions will know which ingredient you are ingesting before each exercise trial (i.e., the double-blind portion of the study). We will also randomize the order of which supplement plus placebo or placebo alone you will ingest so neither you nor the research assistant testing will know this either. The cross-over part of the study is that you will complete 2 testing sessions to assess some physical performance variables (grip strength, jump height and power, and anaerobic energy system power output) with one-week of a wash-out period between them. This will allow us to compare the placebo session to the active nutritional supplement plus placebo condition to evaluate if the supplements improve exercise performance acutely.

You will also be asked to fill in a 24-hour food and fluid log for the period before your initial exercise test. Then you will be asked to repeat this food and fluid intake when completing the second session. No caffeine, alcohol, or vigorous exercise will be allowed for the 24-hours prior to each trial.

ELIGIBILITY:
Inclusion Criteria:

* Recreationally physically active individuals will be recruited for the study. In this context it means all participants perform 1-hour of exercise per day over 3-days per week at a minimum for 1-month. All participants will be between the ages of 18-39 years of age.

Exclusion Criteria:

* Exclusion criteria for the study includes: 1) smokers; 2) unhealthy (have cardiovascular, metabolic, neurological, or psychological disease); 3) taking medication for any condition; 4) any known allergy to the supplements of interest (L-arginine or placebo [dextrose]).

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Grip Strength | 5 minutes
  Grip strength measurement in kilograms of force produced on a hand held dynamometer.
Counter movement vertical jump | 3 minutes
  Counter movement vertical jump performance height in centimeters.
Wingate anaerobic cycle ergometer test | 30 seconds
  Maximum pedaling power output for 30 seconds of all-out sprinting on a cycle ergometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Applied Research Centre; Active Living Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No